CLINICAL TRIAL: NCT04736433
Title: Replication of the PARADIGM-HF Heart Failure Trial in Healthcare Claims Data.
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-PARADIGM-HF
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Angiotensin-Converting Enzyme Inhibitors; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACE Inhibitors: Reference group
  Interventions: Drug: ACE inhibitor
- Sacubitril/Valsartan: Exposure group
  Interventions: Drug: Sacubitril/Valsartan

INTERVENTIONS:
Drug: ACE inhibitor — ACE inhibitor dispensing claim is used as the reference
  Groups: ACE Inhibitors
Drug: Sacubitril/Valsartan — Sacubitril/Valsartan dispensing claim is used as the reference
  Groups: Sacubitril/Valsartan

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

All patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of sacubitril/valsartan or a ACEi (cohort entry).

Eligible cohort entry dates:

Market availability of sacubitril/valsartan in the U.S. started on July 7, 2015.

* For Marketscan: July 7, 2015 - December 31, 2018 (end of data availability)
* For Optum: July 7, 2015 - March 31, 2020 (end of data availability)
* For Medicare: July 7, 2015 - December 31, 2017 (end of data availability)

Inclusion Criteria:

* Age 18 years or older
* NYHA functional class II-IV
* LVEF ≤ 35%

AND the following:

* Hospitalization for heart failure within the last 12 months

  * Treatment with a stable dose of an ACE inhibitor or an ARB equivalent to enalapril 10 mg/day for at least 4 weeks before the screening visit; and treatment with a stable dose of a beta-blocker for at least 4 weeks prior to the screening visit, unless contraindicted or not tolerated
* Treatment with a stable dose of an ACE inhibitor or an ARB equivalent to enalapril 10 mg/day for at least 4 weeks before the screening visit

AND the following:

* Treatment with a stable dose of a beta-blocker for at least 4 weeks prior to the screening visit, unless contraindicated or not tolerated

Exclusion Criteria:

* Known history of angioedema
* Requirement for treatment with both ACEIs and ARBs
* Current acute decompensated heart failure (exacerbation of chronic heart failure manifested by signs and symptoms that may require intravenous therapy)
* Symptomatic hypotension and/or a systolic blood pressure <100 mmHg at Visit 1 (screening) or <95 mmHg at Visit 3 or at Visit 5 (randomization)
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 at Visit 1 (screening), Visit 3 (end of enalapril run-in), or Visit 5 (end of LCZ696 run-in and randomization) or >35% decline in eGFR between Visit 1 and Visit 3 or between Visit 1 and Visit 5
* Serum potassium >5.2 mmol/L at Visit 1 (screening) or >5.4 mmol/L at Visit 3 or Visit 5 (randomization)
* Acute coronary syndrome, stroke, transient ischaemic attack, cardiac, carotid, or other major cardiovascular surgery, PCI, or carotid angioplasty within the 3 months prior to Visit 1.
* Implantation of a cardiac resynchronization therapy (CRT) device within 3 months prior Visit 1 or intent to implant a CRT
* History of heart transplant or on a transplant list or with LV assistance device
* History of severe pulmonary disease
* Diagnosis of peripartum- or chemotherapy-induced cardiomyopathy within the 12 months prior to Visit 1
* Documented untreated ventricular arrhythmia with syncopal episodes within the 3 months prior to Visit 1
* Documented ventricular arrhythmia within the 3 months prior to Visit 1

AND the following:

* Syncopal episodes within the 3 months prior to Visit 1

AND the following:

* Untreated ventricular arrhythmia within the 3 months prior to visit 1

OR the following:

* Untreated ventricular arrhythmia within the 3 months prior to visit 1
* Symptomatic bradycardia or second- or third-degree atrioventricular block without a pacemaker
* Presence of haemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to LV dilatation
* Presence of other haemodynamically significant obstructive lesions of the LV outflow tract, including aortic and subaortic stenosis
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs, including, but not limited to, any of the following:
* History of active inflammatory bowel disease during the 12 months before Visit 1

OR the following:

* Active duodenal or gastric ulcers during the 3 months prior to Visit 1

OR the following:

* Evidence of hepatic disease as determined by any one of the following: aspartate aminotransferase or alanine aminotransferase values exceeding 2× upper limit of normal at Visit 1, history of hepatic encephalopathy, history of oesophageal varices, or history of porto-caval shunt

OR the following:

* Current treatment with cholestyramine or colestipol resins
* Presence of any other disease with a life expectancy of 5 years
* Any Ivabradine use -- Approved in April 2015 (same year as Entresto)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group retrospective cohort study design comparing sacubitril/valsartan to ACE inhibitors. Although the trial compared sacubitril/valsartan to enalapril, we expanded the definition of the comparator group to include all ACEi therapies to improve power, since all medications within this class of medication are indicated and guideline recommended for use in heart failure with reduced ejection fraction patients and would be expected to have similar effects on the primary outcome of CV death and HF hospitalization.
  The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of sacubitril/valsartan or a ACEi (cohort entry).
Sampling Method: Probability Sample
Enrollment: 6066 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Composite outcome of death from cardiovascular causes or hospitalization for heart failure | Through study completion (a median of 102-139 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT04736433/Prot_001.pdf